CLINICAL TRIAL: NCT04785963
Title: Effect of Music and Other Audio Recordings for Chronic Pain in Aging Adults: A Randomized Controlled Study
Brief Title: Effect of Music and Other Audio Recordings for Chronic Pain in Aging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Gary R. Elkins, Director of Mind-Body Medicine Research Lab, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1863320-38
Record Dates: First submitted 2021-02-25; First posted 2021-03-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain; Chronic Pain; Sleep; Aging
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Suggestion; Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music with Suggestion (Experimental): Active condition where participants will be provided with recordings of pre-determined music in addition to recorded suggestions instructing the participant on how to listen to the music.
  Interventions: Behavioral: Music with Suggestion
- Music (Active Comparator): Control group where participants will be provided recordings of pre-determined music
  Interventions: Behavioral: Pain Information
- Pain Information (Active Comparator): Non-arts group receiving structured attention and standard care
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music with Suggestion — A nonpharmacological, short-term treatment that poses minimal risk and places very limited burden on patients seems ideal for this population, and music with suggestions is one such treatment option.
  Arms: Music with Suggestion
Behavioral: Pain Information — The comparison condition of informational recordings about chronic pain are structured to account for non-specific effects of general time and attention and to evaluate whether the treatments of music alone, and music in combination with suggestion are effective in the reduction of pain intensity more than an appropriate control group.
  Arms: Music
Behavioral: Music — The comparison condition of the music only is structured to account for the effect of music listening, and to evaluate whether the addition of suggestion optimizes its effectiveness in the reduction of pain intensity.
  Arms: Pain Information

SUMMARY:
The long-range goal is to reduce suffering and establish alternative options for older adults experiencing pain. This is a randomized controlled study examining the effect of music on pain management in older adults.

DETAILED DESCRIPTION:
Study Objectives:

1. Evaluate the efficacy of the music with suggestion intervention for chronic lower back pain in aging adults, with the indication that music with suggestion will significantly decrease subjective measures of pain compared to controls of music without suggestion or an informational recording about chronic pain.
2. Evaluate the efficacy of the music with suggestion intervention for sleep in aging adults, with the indication that music with suggestion will significantly improve subjective measures of sleep compared to controls of music without suggestion or an informational recording about chronic pain.
3. Evaluate the efficacy of the music with suggestion intervention for mood in aging adults, with the indication that music with suggestion will significantly improve subjective measures of mood compared to controls of music without suggestion or an informational recording about chronic pain.

Recruitment Plan

There will be 66 participants who wish to utilize mind-body interventions as treatment for chronic lower back pain.

The individual's eligibility will be determined using an Inclusion/Exclusion Criteria Screening Checklist containing the criteria listed above. If an individual appears to be eligible, he/she will be educated about the study purpose, procedures, and requirements. If the individual is interested in participating, they will sign a consent form, which may be signed through mail, through electronic platforms such as DocuSign, or in-person. The participant will be scheduled for their first formal education session and informed consent will take place during this session. This education session will take place through a video conference platform. All three groups will meet with a research staff member approximately five times (once during the education session and approximately once per week each following week) throughout the duration of the study. These sessions will take place through a video conference platform.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 50 years of age
2. Participant must regularly experience moderate to severe chronic, lower back pain as determined by a self-reported pain rating of ≥ 5 on 11-point numerical rating scale
3. Duration of pain must be ≥ 6 months
4. Participant must be proficient and able to speak, read, and write in English
5. Participant must have access to a computer or mobile device, Internet, and be willing to participate in virtual sessions and use electronic platforms to complete materials

Exclusion Criteria:

1. Presence of any psychiatric condition or symptom that would interfere with participation, specifically active suicidal ideation with intent to harm oneself or active delusional or psychotic thinking
2. History of mental illness (i.e., psychosis, schizophrenia)
3. Non-English speaker
4. Pain classified as neuropathic as detected by the Pain Detect Questionnaire

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Scale | Daily
  Subjective measures of pain intensity, which will be determined using a Pain Intensity Scale. This measure will be completed daily where participants will be asked to rate the intensity of their pain on a scale from 0 (No Pain) to 10 (Very Intense Pain). Higher scores will indicate greater pain intensity.

SECONDARY OUTCOMES:
Pain Suffering Visual Analogue Scale (VAS) | Weekly up to 4 weeks
  To measure pain suffering. Participants will be asked to rate their level of suffering from pain on a 0 (No Suffering) to 10 (Extreme Suffering) scale. Higher scores will indicate greater pain suffering.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form | Weekly up to 4 weeks
  To measure sleep disturbance. This scale measures self-report 1) sleep quality, 2) sleep depth, and 3) restoration associated with sleep. This scale includes 8 items measured on a 5-point scale.
Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression-Short Form | Weekly up to 4 weeks
  To measure depression. This measure assesses self-reported experiences of negative mood, decreased positive affect and decreased engagement over the past 7 days on a 1 (never) to 5 (always) scale. This scale includes 8 items with higher scores indicating greater depressive symptoms.
Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety- Short Form | Weekly up to 4 weeks
  To measure anxiety. This measure assesses self-reported fear, worry, dread, hyperarousal, and somatic symptoms related to arousal over the past 7 days on a 1 (never) to 5 (always) scale. This scale includes 8 items with higher scores indicating greater anxiety symptoms.
Relaxation Visual Analog Scale | Weekly up to 4 weeks
  To measure relaxation. Participants will be asked to rate their level of relaxation on a scale from 0 (Not Relaxed at All) to 10 (Very Relaxed). Higher scores will indicate greater relaxation.
Self-report of medication use | Daily up to 4 weeks
  Medication use measured by participants' daily self-report of medication use.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No